# **ASCEND STUDY PROTOCOL**

ASCEND: ApproacheS to CHC ImplEmeNtation of SDH

Data Collection and Action

NCT03607617

Version: September 27, 2021

This Version Approved by Kaiser Permanente – Northwest IRB on September 30, 2021

### 1. Protocol Title

ASCEND: ApproacheS to CHC implEmeNtation of SDH data collection and action

### 2. Objectives

ASCEND will test strategies for helping community health centers (CHCs) systematically identify and take action on social determinants of health (SDH). This work builds on our NIDDK-funded pilot study (R18DK105463), in which we developed a set of electronic health record (EHR) tools for SDH data collection and summary. These tools were activated in 440 primary care CHCs nationwide in June 2016. We propose to act on this unique opportunity to study: (i) SDH data collection / action in CHCs in 19 states; and (ii) the effectiveness of a set of implementation strategies at supporting CHCs in integrating SDH data collection and action into workflows and DM risk management care plans.

Note: The SDH intervention includes strategies to help CHC's systematically (i) collect SDH data in standard workflows using EHR tools and (ii) integrate SDH data from flowsheets into care plans (e.g., making referrals to social services; adapting treatment plans) for adults with / at risk for DM. The study team will provide intensive implementation support (in the form of technical assistance and training materials) to study CHCs.

Focusing on DM risk management and obesity prevention outcomes in adult patients, we will:

Aim 1. Conduct a mixed methods formative evaluation of SDH data collection uptake among CHCs that had SDH data tools activated in their EHR in June 2016. (Quantitative data will come from all 440 CHCs' shared EHR, qualitative data from up to 12 CHCs purposively recruited from this pool). Identify patterns of SDH data collection in these diverse CHCs, and clinic-level factors associated with variation in SDH data collection rates. Use results to fine-tune the SDH Action Plan intervention's strategies for helping CHCs systematically: (i) collect SDH data in standard workflows, and (ii) integrate SDH data into care plans (e.g., making referrals to social services; adapting treatment plans) for adults with / at risk for DM.

Aim 2. Conduct a pragmatic, stepped-wedge, cluster-randomized trial in 30 CHCs. The CHCs will be randomized to one of six wedges, with staggered timing. CHCs in each wedge will receive intensive implementation support (the SDH Action Plan). This scalable intervention includes both comprehensive technical assistance and training materials designed to help CHCs plan for and implement SDH data collection / action, and six months of remote access to an 'SDH Implementation Team' that will tailor implementation support to each CHC's needs, with an emphasis on the Building Blocks of Primary Care. (The SDH Action Plan will be fine-tuned based on Aim 1 results, and a baseline survey of the study CHCs.)

**Aim 3:** Conduct a process evaluation of whether and how the SDH Action Plan intervention improves: (i) SDH data collection in CHC workflows; (ii) integration of SDH data into DM risk management care; and (iii) clinical measures associated with effective DM risk management (controlled blood pressure, HbA1c, BMI, lipids, etc.; up-to-date preventive care). *H3a:* Intervention CHCs will have significantly greater increases in (i) SDH data collection, and (ii) actions taken to address SDH needs, compared to control CHCs. *H3b:* Patients at intervention CHCs for whom SDH data are collected will have significant improvements in DM / obesity risk management / receipt of related preventive care, compared to those at control CHCs.

### 3. Background

Research is needed on how to help community health centers (CHCs) start collecting and taking action on patient-reported SDH data. CHCs serve our nation's most vulnerable patients, whose DM prevalence and risk (notably, obesity rates) are higher than the general population's, and whose health is particularly impacted by SDH. At present, CHC staff may seek to identify whether SDH are impacting a patient's ability to act on care recommendations for DM prevention / management, and / or whether DM care plans should be modified to address these SDH. However, such efforts are typically ad-hoc, and rarely involve structured EHR data as recommended by public health leaders. There is a pressing need to identify barriers to CHCs

systematically screening for and acting on SDH using EHR-based tools, and to determine whether implementation strategies that support other practice changes can effectively address these barriers.

We propose to test a SDH intervention (also referred to as a set of strategies) for helping CHCs routinely identify and take action on the SDH-related needs of patients with / at risk for DM. The proposed work builds on our pilot study called Assess & Do (R18DK105463), which used a stakeholder-driven process to develop EHR-based SDH data collection / summary tools for CHCs. The ASESSS&DO study is Pro00005883 within the IRB system.

Please refer the end of this document for a bibliography.

### 4. Study Design

ASCEND is a pragmatic trial which assesses whether / how an implementation support intervention impacts SDH data collection / action and DM risk management, in 30 CHCs. We will tailor the support provided to meet each CHC's needs, while ensuring that any support could be replicated in usual care, so that study findings are useful to healthcare decision-makers. Our intervention, delivered in routine care settings, addresses recent calls to study methods for adapting change management strategies to meet setting-specific needs.

We propose a mixed methods, stepped-wedge, cluster-randomized trial to assess the effectiveness of a set of evidence-based, pragmatic approaches to helping CHCs implement SDH data collection / action, in care for adults with / at risk for DM / obesity.

We hypothesize that intervention CHCs will have significantly greater increases in (i) SDH data collection, and (ii) actions taken to address SDH needs, compared to control CHCs. We also hypothesize that patients at intervention CHCs for whom SDH data are collected will have significant improvements in DM / obesity risk management / receipt of related preventive care, compared to those at control CHCs.

### 5. Study Population

### a. Number of Subjects

First, we will pull data on CHCs from the OCHIN membership database; OCHIN has agreements with their member CHCs for such data extraction and analysis.

Then, we will recruit CHCs from this pool based on high adoption rates at baseline (N=no more than 12). From these 10-12 CHCs, we will interview up to 6 CHC staff (total N=72) as part of formative data collection efforts.

Next, we will recruit up to 31 CHCs, and conduct block randomization to one of six study wedges for staggered receipt of the SDH Action Plan (N= up to 31). Thus, a maximum of 43 CHCs will participate in the study; although some CHCs that participate in the formative interviews may also opt to be included in the study phase, meaning we may not recruit 42 unique CHCs.

We will ask CHC champions in the 31 CHCs to oversee completion of a baseline survey before the SDH Action Plan intervention is implemented. The subsequent process evaluation will include a card study with selected providers at each clinic, and content analysis of interactions between the implementation support team and CHC staff.

Total maximum participants for each aspect of the study

CHCs: up to 43 total

### CHC staff:

- Phone /in-person interviews: 72 (cross-section of staff)
- Baseline surveys: ~ up to 50 (project champions at each clinic)
- Card study: up to 62 (primary care providers)

 Content analysis of OCHIN's SDH implementation team interactions with study CHC staff (text data from recorded webinars, emails, online discussions between OCHIN implementation team and CHCs)

### b. Inclusion and Exclusion Criteria

### **Quantitative Data**

### **Inclusion Criteria:**

- Any patient who had an encounter at an OCHIN member facility between June 24, 2016 (when tools went live) and December 31, 2022.
- Pregnant women
- Children
- May include some subjects with mental health conditions of various types; however, it is
  important to systematically address high DM /obesity risk in this population, because such
  patients may be at risk for elevated high DM /obesity risk and have often been excluded or
  underrepresented in previous research studies.
- Decisionally/cognitively impaired
- Economically/educationally disadvantaged
- Non-English Speakers
- Elderly

Note: Social determinants of health (SDH) information may be incidentally collected using the tools of this project at the discretion of the clinics. The project is designed to allow them to use the SDH tools in a way that best fits the individual clinics' needs. This study is looking specifically at the impact of SDHs on diabetes, however SDHs are important factors for many aspects of clinical care. Based on previous work around SDHs, clinics may collect SDH information for children or pregnant women in their practice as a tool to guide their care. As a result, the inclusion of SDH data for all patients that have been screen for SDH needs is important for the project to understand the extent of the tool's use across their entire patient population. The inclusion of pregnant women will be limited by the extent to which the participating clinics administer the tool to their patient population but will not be specifically targeted as a participation criterion. However, aggregated descriptive analyses will include an indicator for pregnancy to understand the frequency and utility for use of these tools in this population. All data will be housed securely in the EMR and only reported at an aggregate level. They will be part of the limited dataset for analyses and protected according to the data security procedures described in this protocol.

# Exclusion Criteria:

- Neonates of uncertain viability or nonviable neonates (up to 28 days post birth)
- Prisoners

*Note:* The investigators are not enrolling patients for this clinic-randomized study, but rather studying the uptake and impact of a set of EHR-based clinical decision support tools into regular care at the participating clinics. In this clinic-randomized trial, the intervention / randomization occurs at the clinic level. The intervention targets clinic processes that are part of the regular care patients receive and will not require special visits.

### **Qualitative Data**

### Inclusion Criteria:

• CHC staff: Employees who are specifically and intentionally targeted to be included in this study population because of their workplace and/or employee status

### **Exclusion Criteria:**

None

### c. Vulnerable Populations

As mentioned above, we will exclude the following vulnerable populations from the study:

- Neonates of uncertain viability or nonviable neonates (up to 28 days post birth)
- Prisoners: Prisoners are excluded or not anticipated to become study subjects

### d. Setting

OCHIN, Inc., is a non-profit, community-based health center-controlled network. Its members (>480 CHCs, in 19 states) share characteristics of other CHCs, so results will be generalizable to many CHCs. As the nation's largest CHC network with a single EHR system, OCHIN pioneered the development of EHR tools for CHCs. OCHIN's member CHCs share a single Epic© EHR, which is unduplicated, centrally maintained, and network-wide. Data are standardized and quality-checked: thus, validated data are already linked between all study sites.

OCHIN will rely on CHR's IRB for IRB review. As with previous studies, OCHIN will submit their cede letter after we are funded. We anticipate that OHSU (Dr. Miguel Marino; lead biostatistician with expertise in complex biostatistics, cluster-randomized, stepped-wedge design) and University of Massachusetts Medical School (Dr. Arvin Garg; co-investigator with expertise in SDH data collection in pediatric care) will cede IRB approval as well.

### e. Recruitment Methods

This study has no formal patient recruitment, as 'participants' will be the CHCs that volunteer to take part in the study. Patients will interact with clinicians as they normally would; the intervention will give clinicians tools for managing patient data during encounters and panel management. We will collect qualitative data from CHC staff as described in the proposal. Below is a summary of recruitment.

CHCs will be recruited by an OCHIN research associate. Materials used for recruitment of clinics will include a participation information sheet, a slide deck with information about study participation, and a recruitment card with a brief description of what we are offering clinics.

### CHC staff:

- Phone / in-person interviews: up to 72 (cross-section of staff) will be recruited by OCHIN staff, in partnership with CHR's qualitative team
- Baseline surveys: ~50 (project champions at each clinic)
- Card study: up to 62 (primary care providers)
- Content analysis of OCHIN's SDH implementation team interactions with study CHC staff (text data from recorded webinars, emails, online discussions between OCHIN implementation team and CHCs)

### f. Consent Process

We are requesting a waiver of informed consent for all data collection activities; details below. ASCEND is a pragmatic trial and obtaining signed consent would unnaturally restrict our study sample, diminishing the external validity of our findings. The project is promoting standard clinical care and quality improvement in the CHC setting. We believe that a waiver of informed consent will not adversely

impact clinic staff. For this study, we are simply overseeing CHC interactions with OCHIN about their workflow implementation. We are not asking for any personal information from staff or patients. It would be impractical to ask for consent as anybody in the clinic could ask for OCHIN support over these 6 months, and we'd inevitably miss someone. No data will be collected from or about patients.

**Formative: Semi-structured phone or in-person interviews with CHC staff:** We will ask for verbal consent prior to conducting the interviews. We have submitted a copy of the ASCEND Study Fact Sheet and Interview guide with this IRB application. This Fact Sheet includes the key elements of consent.

### 6. Study Procedures

### Aim 1

### Clinic Recruitment

• Up to 12 CHCs will be recruited from OCHIN's pool of clinics to participate in semi-structured interviews.

## **Mixed Methods Formative Evaluation**

- The qualitative team will conduct semi-structured interview to explore barriers / facilitators to EHR-based SDH data collection / use in DM-related care, with a focus on contextual factors. At each CHC, we will conduct ≈6 phone / web interviews with a cross-section of staff including, as appropriate, medical directors, primary care providers (MD, PA, NP) / team members (MA, RN), and staff members responsible for QI (clinic managers, care managers) / ad-hoc SDH management (e.g., social workers). We will ask how SDH information is now used to inform care, challenges to collecting / using SDH data, experiences with the EHR's SDH data tools, and how to facilitate SDH data collection / action. Verbal consent will be obtained pre-interview.
- The quantitative team will collect baseline data from 6/24/16-12/31/17 for the 440 CHCs that share OCHIN's EHR. We will measure clinic-level SDH data collection rates as percentage of adult patients seen in 6/24/16-12/31/17 for whom patient-reported SDH data from the IOM's list are recorded, on a monthly basis. We will assess variation in rates of SDH data collection and identify clinic-level factors associated with this variation, using standard statistical methods. The distribution of the outcomes of interest and eligible population will be examined before selecting an analysis model; specific models will be refined iteratively, guided by the hypotheses and conceptual model.

### Fine-tune the SDH Action Plan

• Results from the formative evaluation (semi-structured interview and baseline data analyses) will be used to fine-tune the SDH Action Plan.

### Aim 2

### Clinic Recruitment and Randomization

• CHCs will be recruited in two separate waves for the pragmatic trial. Wave 1 (wedges 1, 2, and 3) will be recruited prior to the start of wedge 1. Wave two (wedges 4,5,6) will be recruited roughly 1 year later, prior to the start of wedge 4. Each wave of CHCs will be block randomized by baseline rates of SDH data collection.

Pragmatic, Stepped-wedge Trial

- The implementation support team will provide tailored implementation support for SDH data collection / action to each CHC's needs for six months (one wedge at a time).
- CHC Staff Baseline Survey: Using the 'Building Blocks of Primary Care' (BBPC) model, we will assess the study CHCs' baseline status of four foundational components/'building blocks': (1) Engaged leadership; (2) Data-driven improvement using EHRs; (3) Empanelment; and (4) Teambased care. The survey will be completed by project champion at each clinic. We will send a survey asking about the CHCs' structural characteristics (payment, staffing, etc.), external policies and incentives that might have an impact, and other potentially impactful organizational characteristics not identifiable in EHR data, OCHIN member records, or the other baseline data. This information will help us understand the impact adoption of SDH data collection / action.
- Baseline EHR data: Aim 1 baseline data will be used to identify baseline SDH data collection / action in the trial CHCs, and to indicate which of these CHCs may need targeted assistance.
   These data will be pulled in the month prior to wedge implementation.
- Card study (short provider survey): Two providers at each CHC will be asked to complete a brief survey ("card") within the EHR following selected patient encounters. Patient encounters will be selected based on the clinic's specified target population for SDH screening. These card studies will be administered over approximately 3 weeks in month 5 of each study wedge. OCHIN will identify two providers that see the majority of their clinics' specified target population and work with the clinic project champion to recruit the providers to participate in this survey. If clinics do not identify a target population, then OCHIN or the study CHC will identify the two providers who screen the most patients for SDH or identify two providers who see the most patients. Each provider will be asked to complete one card immediately after an office and / or telehealth encounter with a patient. PCPs will access the card study questions via a link built into the EHR. Responses will be pulled from the Clarity database by the OCHIN analyst. Each "card" will be associated with the following characteristics: responses from provider for card study questions, SDH screening reported, SDH need(s) documented, reason for visit, patient demographics, and provider and site information.

The card study questions will ask questions such as: (1) Whether / how SDH data informed clinical decisions / actions; (2) How the SDH data was obtained (e.g., via the EHR tools); (3) Whether any desired SDH data were unavailable; and (4) Estimated time spent looking up SDH data. Answers will be fixed-choice with an "other" option and space for free text. No PHI will be captured, and provider answers will not be stored in patients' charts.

The qualitative team will present a card study information sheet to the clinics in month 4 of each wedge.

- Member checking survey: The qualitative team will prepare clinic specific paragraphs of our learnings, barriers, and facilitators. We will ask up to 2 clinic champions per clinic to review this paragraph and answer questions about their SDH screening post-end wedge. The survey will be sent out via email within the body of the email or using a survey platform link. The study team will send a reminder email within one week of sending out the survey.
- Content analysis of CHC / implementation support team interactions: Prior to study
  participation, we will notify CHC staff that their exchanges with the implementation support
  team will be analyzed for research purposes. Staff participation will serve as implied consent.
  There is no contact with patients. We are observing to identify barriers and facilitators to
  implementation (akin to document review, which we have used in previous studies for email
  exchanges, clinic meeting minutes, etc.).

All exchanges with study CHCs will be used in content analysis; calls and webinars will be recorded (with permission) and transcribed; emails / online discussions will be collected. The OCHIN and CHR teams may incidentally view and record PHI while helping clinics implement the SDH EHR tools as part of the webinar sessions. Recording PHI is not intended to contribute to the research question and any PHI inadvertently captured would be deleted before the data is used in analysis.

When each wedge ends, the qualitative team will record a debrief session with the SDH Implementation Team to capture their understanding of implementation at each CHC in that wedge. We will also collect 'trouble-tickets' about the SDH tools submitted to OCHIN's member support system.

Assess the relationship between clinic context and implementation strategy adaptation: We will
track context and implementation strategies including planned, unplanned, enacted, and
adapted strategies and justifications for strategy adaptation. We will use a comparative case
study approach to compare strategies between sites, document adaptations, and explore
preliminary patterns of association between context, strategies, and outcomes.

We will synthesize meeting notes, transcripts, and email which document interactions between the research team and each clinic, internal planning meetings between research team members, and clinics' use of intervention guidance and decisions tools.

#### Aim 3

### Mixed methods process evaluation

- We will analyze the quantitative data and qualitative data to understand whether and how the SDH Action Plan intervention improves:
  - 1. SDH data collection in CHC workflows;
  - 2. integration of SDH data into DM risk management care; and
  - 3. clinical measures associated with effective DM risk management (controlled blood pressure, HbA1c, BMI, lipids, etc.; up-to-date preventive care).
- We will also analyze the quantitative and qualitative data to:
  - Examine the impact of screening domain, patient characteristics, clinical encounter characteristics, and clinic factors and on accepting on refusing help to address a social need.
  - Characterize variability in food insecurity and other social risk screening implementation before and during the COVID-19 pandemic, with an emphasis on screening during telehealth encounters, using multilevel data.
  - Identify barriers and facilitators to food insecurity and other social risk screening implementation before and during the pandemic, with an emphasis on screening during telehealth encounters

### **Data Collection**

### Quantitative data points

• Aim 1 data points - We will collect baseline data from 6/24/16-12/31/17 for the 440 CHCs that share OCHIN's EHR. We have extracted similar EHR data in prior research. We will measure

clinic-level SDH data collection rates as percentage of adult patients seen in 6/24/16-12/31/17 for whom patient-reported SDH data from the IOM's list are recorded, on a monthly basis. We will assess variation in rates of SDH data collection and identify clinic-level factors associated with this variation, using standard statistical methods. The distribution of the outcomes of interest and eligible population will be examined before selecting an analysis model; specific models will be refined iteratively, guided by the hypotheses and conceptual model. Results from these analyses will inform clinic recruitment and fine-tuning of the intervention as described below.

- Aim 2 & 3 data points -
  - Monthly rate of targeted patients for whom SDH data are documented in the EHR.
  - Monthly rate of patients for whom an SDH-related referral is made (exclude if 'patient declined referral' is documented).
  - Control of DM risk management biomarkers: (i) BP control (<140/80 mmHg); (ii) A1c control (<7.0%); (iii) BMI <30; (iv) LDL control (I<100 mg/dL).</li>
  - Rates of incident comorbidities, e.g. retinopathy, nephropathy, neuropathy (among patients with DM).
  - Rate of patients up-to-date on DM key tests (e.g. lipid panel annually, HbA1c within 6 months..)

### **Qualitative data points**

- Aim 1: Formative, semi-structured interviews.
- Aim 2 & 3: Baseline survey at study clinics, card study (short provider survey), exchanges between CHC staff and implementation support team (can include, but is not limited to: emails, webinar recordings, meeting notes, ASCEND SDH Toolkit, etc.), and the member checking survey.

## 7. Data Analysis

### a. Analysis Plan

# Quantitative data analysis plan

All quantitative analyses will be led by co-I Dr. Marino from OHSU. This stepped-wedge cluster randomized trial will evaluate the impact of the proposed intervention on our dependent variables (see Table 6 in proposal): adoption of SDH data collection / action, and impact of this adoption on DM risk management. Outcomes will be measured monthly in all clinics at every period, so that each wedge provides data points in both control and intervention conditions. Practices in each wedge will be block-randomized by baseline rates of SDH data collection to balance SDH collection adoption across wedges. The main goal of this trial is to establish whether the intervention is effective and to what degree. Our evaluation includes a rigorous design so we may attribute positive findings to the intervention. To compare the effect of the intervention with usual practices on SDH outcome measures in a stepped-wedge design, we will utilize Generalized Linear Mixed Models (GLMMs).

Quantitative data analyses will use elements from The Limited Data Set. Data elements will contain the following variables and/or variables that have been derived from these variables (such as counts, means, etc.) ("Data Elements") between June 24, 2016 and December 31, 2022:

| Category | Examples include, but are not limited to: |
|---|---|
| Demographics | Patient ID, sex, date of birth, race, ethnicity, primary language, annual |
| | income, FPL, primary payor, state of residence, urban/rural |
| Encounter | Encounter ID, patient ID, admit date, provider ID, facility location, |
| | encounter type, facility id, admitting source, primary payor, site ID |
| Diagnosis | Diagnosis ID, patient ID, encounter ID, encounter type, admit date, provide |
| | ID, diagnosis, diagnosis type, diagnosis source, site ID, comorbidity index |
| | score |
| Procedures | Procedures ID, patient ID, encounter ID, encounter type, provider ID, |
| | procedure date, procedure code, procedure type, procedure source, site ID |
| Vital | Vital ID, patient ID, encounter ID, measure date, measure time, vital source, |
| | height, weight, diastolic blood pressure, systolic blood pressure, original |
| | BMI, blood pressure position, smoking, tobacco, tobacco type, site ID |
| Lab Result CM | Lab result cm ID, patient ID, encounter ID, lab name, specimen source, raw |
| | lab name, lab loinc, result location, lab procedure, lab procedure type, lab |
| | order date, result date, result quality, result number, result modifier, result |
| | unit, norm range low, norm range high, norm modifier high, abnormal |
| | result indicator, site ID |
| Condition | Condition ID, patient ID, encounter ID, report date, onset date, resolve |
| | date, condition status, condition, condition type, condition source, site ID |
| Prescribing | Prescribing ID, patient ID, encounter ID, ID provider ID, Rx order date, Rx |
| | start date, Rx end date, Rx quantity, Rx refills, Rx days supply, Rx frequency, |
| | Rx basis, Rx norm concept identifier, site ID |
| Clinic Characteristics | Patient portal use, years on EHR, AHC participation |
| Provider | Sex, credentials, specialty, years practicing at clinic, number of visits, SDH |
| Characteristics | tool use |
| Social Determinants of | SDH need, education, financial resource strain, housing insecurity, food |
| Health | insecurity, intimate partner violence, inadequate physical activity, social |
| | isolation, stress, request for help |

Additional quantitative data analyses will include assessing SDH data collection / action, overall and among the subset of clinics that are both OCHIN-member clinics and part of the Accountable Health Communities (AHC) study at OHSU, as well as all OCHIN member CHCs during a time when federal initiatives are emphasizing this change. We will track SDH data collection rates in these CHCs over study years 1-4, in descriptive analyses.

We will also use a generalized estimating equation (GEE) approach to assess factors associated with patients' acceptance of a resource to address an identified social need (see model specification below). Acceptance of help will be calculated using the proportion of patients who screened positive for one or more social need who accept a help to address that need. GEE produces a population average effect that accounts for group-level correlation and is appropriate for repeated or correlated observations. To account for the likely correlation between patients within a clinic, the model will include clustering at the clinic level. GEE takes into account the specified correlation structure while selecting the final parameter estimates and generally controls for clustering more effectively than using post-processing adjustment. We will test exchangeable and unstructured correlations structures and compare models using Quasi-Likelihood AIC (QIC) test. We will select the model with the lower QIC value. Using the

preferred model, we will assess predictors of positive screening including screening domain, patient characteristics, encounter characteristics, and clinic characteristics.

 $Y_i$  Patient acceptance =  $\beta_0 + \beta_1 X_i$ Screening domain +  $\beta_2 X_i$ Patient characteristics +  $\beta_3 X_i$ Encounter characteristics +  $\beta_4 X_i$  Clinic characteristics +  $u_i$ 

To characterize variability in food insecurity and other social risk screening implementation before and during the COVID-19 pandemic, we will use a multilevel mixed-effects model to predict implementation of screening based on site, provider, patient, and visit characteristics. Variables will include urbanicity at the site level; profession at the provider level; race/ethnicity, age, and number of diet-related chronic conditions at the patient level; and location (in-person v. telehealth) at the visit level.

### Qualitative data analysis plan

Data from each case will be 'merged' for analysis, then compared within and across clinics to confirm, expand on, or challenge each site's finding. Data collection and analysis will be parallel and iterative; analysis will begin at the end of the first wedge and continue as data from each wedge is collected. A grounded theory approach and immersion-crystallization process will be used to identify data themes and patterns.

Qualitative data analyses for the card study will use elements from the below data set. Data elements will include, but are not limited to the following variables:

| Category | Description and Variable Name |
|---|---|
| Provider | Sex, credentials, specialty, years practicing at clinic, number of visits, SDH |
| Characteristics | tool use |
| Encounter characteristics | Encounter date, type, reason for visit |
| Card study responses | What factors influenced the care you provided, how did you know the patient's SDH information, How long did it take to look up the patient's SDH information, how much did SDH influence your clinical decisions |
| Patient-level SDH | SDH need, education, financial resource strain, housing insecurity, food insecurity, intimate partner violence, inadequate physical activity, social isolation, stress, request for help |

Card study response data will be summarized by provider, clinic, and wedge. Analyses will be Ns and percentages of each survey item response and descriptive patient demographic data for the patients whose encounters were selected for inclusion in the card study (e.g., patient sex, age category, race/ethnicity, preferred language, and whether they had any discrete SDH screening data recorded in the EHR).

We will assess the relationship between clinic context and implementation strategy adaptation, we will code implementation strategies and barriers deductively and using ERIC and CFIR respectively and inductively based on themes that emerge from the data. We will incorporate

additional categories proposed based on the application of ERIC categories across several large interventions and analyze data as comparative case studies.

We will also analyze clinic communications using a constant-comparative approach and merge that with quantitative data in joint display tables to characterize variability in food insecurity. An implementation framework will be used to develop a model of facilitators and barriers to food insecurity screening.

### b. Sharing of Results with Subjects

The study results will not be shared with subjects. This study does not carry the risk of incidental findings. This study does not involve laboratory results.

### c. Data and Specimen Banking

Not applicable.

### 8. Privacy, Confidentiality, and Data Security

### Quantitative data management, sharing and protection:

Datasets will be created with data from OCHIN's web server and data shared by OHSU for the AHC-participating clinics, imported into SAS, and securely maintained at OCHIN. Data will be extracted for all target patients seen in study CHCs and stored (limited data set) in a secure repository. Data from subsequent encounters is stored and linked to the same patient. Identified patient data will be transferred from OHSU (ORPRN) for the subset of patients seen in OCHIN+AHC clinic sites; these data will include patient identifiers sufficient to match them to their EHR record in the OCHIN system (e.g., name, date of birth, medical record number), as well as SDH screening data necessary for analysis. After matching is conducted, all PHI will be stripped from these datasets and will not be accessed for analysis or transferred back to OHSU as part of Limited Data Sets for analysis.

OCHIN and CHR have expertise in high-quality and secure data management, project operations, and multisite research collaborations. Data structures will remove personal identifiers. Analyses will be done in SAS® v9 or higher. Limited data sets will be shared between OCHIN, OHSU, UNC, and WSU. Please note that OCHIN will send the same final limited dataset to OHSU and WSU. Limited data sets will be password protected for transfer and exchanged via a secure data transfer method. Quantitative data will be securely stored on Dropbox or on an institutional server. Only aggregate EHR data will be shared outside of the study team.

Qualitative data management, sharing and protection: Qualitative data will be securely stored at CHR, OCHIN, UNC, and WSU. All data work will be done on password-protected workstations, in a secure environment (HIPAA-compliant). Data will be catalogued within 1 week of collection, and field notes within 24 hours.

- Interviews will be recorded and professionally transcribed by an outside vendor (with who KPCHR and OCHIN have a Business Agreement with). Recordings will be sent via secure file transfer (SFT) to the transcriptionist.
- Online meeting software recordings (e.g. Zoom or Microsoft Teams) of the monthly webinars will be sent from OCHIN to CHR via SFT, encrypted email, secure site, or Box. Recordings will be sent via

secure file transfer to an approved transcriptionist with whom the study team has an established BAA. The transcriptionist will be instructed to delete any identifiable patient information in the transcript (e.g., [\*Name\*]) and to delete the recording once the transcription is complete. Recordings have the *potential* to contain PHI as a result of the Epic environment that may be used in SDH tool demonstration; transcripts will NOT contain any PHI and PHI will not be used in analysis. The transcript will be sent back to the qualitative study team via secure file transfer (access to the secure file transfer site will be limited to appropriate members of the research team); recordings and transcripts will be stored securely at both CHR, OCHIN, UNC, and WSU. Transcripts will be entered into QSR NVivo or Dedoose. Recordings will be deleted at the end of the study.

 Card study data will be sent via secure site, encrypted email, Secure File Transfer or Box between OCHIN and CHR.

All qualitative data work will be done on password-protected workstations, in a secure environment (HIPAA-compliant). At CHR, only study team members have access to the saved data. At OCHIN, access to study data is limited to the research department. At UNC and WSU, access is limited to study team members. Data files will be password protected for transfer; data sharing agreements / protections will be established as necessary.

Other qualitative data will be entered into QSR NVivo and Dedoose; data files will be password protected; data sharing agreements / protections will be set as necessary; transfers will use a secure website or encrypted email.

<u>Confidentiality measures:</u> All research staff at CHR, OCHIN, OHSU, and WSU who handle data sign confidentiality pledges and receive IRB and HIPAA training/certification.

<u>Security measures:</u> Multiple measures are in place to ensure security of PHI. Data transfer to and from the EHR (at OCHIN), and the web display (accessed at OCHIN member CHCs) uses a Simple Object Access Protocol (SOAP) with Secure Sockets Layer (SSL) encryption over a Hypertext Transfer Protocol Secure (HTTPS) computer network.

### 9. Provisions to Monitor the Data to Ensure the Safety of Subjects

This study involves data from OCHIN's network of safety net clinics, 42 of which will be recruited for formal study participation. All EHR data from OCHIN clinics are stored at OCHIN. Each clinic has business use agreements with OCHIN to handle and manage PHI from their clinical data. EHR data will be linked using OCHIN's unique patient identification codes, in order to create clinic-level aggregate data and a limited data set.

All data sources will be linked into a secure relational database at OCHIN. The de-identification process replaces the original identifiers on sensitive or confidential fields with arbitrary pseudo-identifiers. Access to the "crosswalk" tables that contain mappings of original- to pseudo-identifiers is limited to authorized OCHIN staff; crosswalk tables will not be shared with OHSU or CHR. We will de-identify the following fields:

- Patient ID
- Provider ID
- Encounter ID

Data analysis will be conducted at OCHIN, OHSU, UNC, and WSU. If necessary, to share PHI, we will use a secure data transfer method (e.g., sFTP) with access limited to appropriate members of the research team. IRB and HIPAA approval will be obtained for all study steps. CHR, OHSU and OCHIN have expertise in high-

quality data and secure management and project operations and multisite research collaborations. Data structures are typically designed to separate personal identifiers from other critical data, further enhancing protections.

CHR, OHSU, and OCHIN standards meet or exceed requirements for patient data safety established in the federal HIPAA guidelines. Data structures will derive from the data confidentiality, security, and privacy standards that CHR, OCHIN, and OHSU have in place to meet or exceed all current HIPAA requirements. Quality control will begin with real-time, inter-field checks in the data at OCHIN. Additional back-end checks (for missing data and logical inconsistencies) will be conducted to ensure the highest standards of data reliability. We will examine the distribution and measurement properties of variables before making final decisions about analyses.

### 10. Risks and Benefits

### a. Risks to Subjects

The ASCEND study poses minimal risk. We do not anticipate any physical, psychological, social, legal or economic risks.

### b. Potential Benefits to Subjects

<u>Overall benefits:</u> This research has the potential to provide valuable information on how best to support uptake of standardized collection of patients' SDH data using EHR-based tools, and integration of SDH data into DM / obesity risk management in CHCs.

Quantitative: Patients at the study CHCs will have no defined personal benefit from this project.

<u>Qualitative:</u> Care team members at the study CHCs will have no defined benefits from participating in this project. However, the intervention is designed to optimize identification and management of adult subjects with elevated DM risk. Some providers exposed to this potentially useful CDS may use it to improve their clinical care during the study or after.

### 11. Costs to Participants

CHC patients: There are no new costs to patients as a result of this study; however they will continue to pay for co-pays, routine treatment costs, etc. as part of normal care at their CHC.

CHC staff: There are no costs to staff as a result of this study; other than time spent during interviews and observations.

### 12. Compensation to Participants

CHCs: During Year 1, the recruited CHCs (N=up to 12) will receive an impact fee in the amount of \$300 for participation in formative data collection.

CHC patients: None

CHC staff: During Years 1-4, CHC staff will receive a gift card in the amount of \$25 or \$50 for participation in the interviews and the card study (short de-identified provider survey).

### **Resources Available**

No special resources or expertise are required to conduct this study.

### 13. Drugs or Devices

Not applicable.

### 14. Multi-Site Coordination

CHR will act as the coordinating center for this study. We will ensure that:

- All sites have the most current version of the protocol, consent document, and HIPAA authorization.
- All required approvals have been obtained at each site (including approval by the site's IRB of record).
- All modifications have been communicated to sites and approved (including approval by the site's IRB of record) before the modification is implemented.
- All engaged participating sites will safeguard data as required by local information security policies.
- All local site investigators conduct the study appropriately.
- All non-compliance with the study protocol or applicable requirements will be reported in accordance with local policy.
- Communication of problems, interim results, and study closure.

### 15. Community-Based Participatory Research

This study has system-level support: OCHIN's leadership strongly supports SDH data collection in its member CHCs, which aligns with OCHIN's ongoing efforts to improve care and outcomes in CHCs via EHR-based strategies. In all study steps, the study team will engage OCHIN's operational leadership (including co-I Karen Parr, a CHC clinician and informaticist). We will also engage OCHIN CHC clinicians via existing communication structures. OCHIN has a long history of engaging stakeholders in all system-wide efforts; CHC clinicians serve on standing committees that direct all changes made to OCHIN's EHR.

### References

- (1) Hill J, Nielsen M, Fox MH. Understanding the social factors that contribute to diabetes: a means to informing health care and social policies for the chronically ill. *Perm J.* 2013;17:67-72.
- (2) Clark ML, Utz SW. Social determinants of type 2 diabetes and health in the United States. *World J Diabetes*. 2014;5:296-304.
- (3) Behforouz HL, Drain PK, Rhatigan JJ. Rethinking the social history. *N Engl J Med.* 2014;371:1277-1279.
- (4) Hughes LS. Social Determinants of Health and Primary Care: Intentionality Is Key to the Data We Collect and the Interventions We Pursue. *J Am Board Fam Med.* 2016;29:297-300.
- (5) US Department of Health & Human Services (DHHS). *Healthy People 2010, 2nd Edition.* Washington, DC: US Government Printing Office.; 2000.
- (6) Gold R, DeVoe J, Shah A, Chauvie S. Insurance continuity and receipt of diabetes preventive care in a network of federally qualified health centers. *Med Care*. 2009;47:431-439.
- (7) Gold R, DeVoe JE, McIntire PJ, Puro JE, Chauvie SL, Shah AR. Receipt of diabetes preventive care among safety net patients associated with differing levels of insurance coverage. *J Am Board Fam Med*. 2012;25:42-49.
- (8) Social disadvantage linked to diabetes through chronic inflammation. BMJ. 2013;347:f4368.
- (9) Hsu CC, Lee CH, Wahlqvist ML, et al. Poverty increases type 2 diabetes incidence and inequality of care despite universal health coverage. *Diabetes Care*. 2012;35:2286-2292.
- (10) Jackson CA, Jones NR, Walker JJ, et al. Area-based socioeconomic status, type 2 diabetes and cardiovascular mortality in Scotland. *Diabetologia*. 2012;55:2938-2945.
- (11) Lipton RB, Liao Y, Cao G, Cooper RS, McGee D. Determinants of incident non-insulin-dependent diabetes mellitus among blacks and whites in a national sample. The NHANES I Epidemiologic Follow-up Study. *Am J Epidemiol*. 1993;138:826-839.
- (12) Lysy Z, Booth GL, Shah BR, Austin PC, Luo J, Lipscombe LL. The impact of income on the incidence of diabetes: a population-based study. *Diabetes Res Clin Pract*. 2013;99:372-379.
- (13) Muller G, Kluttig A, Greiser KH, et al. Regional and neighborhood disparities in the odds of type 2 diabetes: results from 5 population-based studies in Germany (DIAB-CORE consortium). *Am J Epidemiol*. 2013;178:221-230.
- (14) Sacerdote C, Ricceri F, Rolandsson O, et al. Lower educational level is a predictor of incident type 2 diabetes in European countries: the EPIC-InterAct study. *Int J Epidemiol*. 2012;41:1162-1173.
- (15) Stringhini S, Sabia S, Shipley M, et al. Association of socioeconomic position with health behaviors and mortality. *JAMA*. 2010;303:1159-1166.
- (16) Espelt A, Kunst AE, Palencia L, Gnavi R, Borrell C. Twenty years of socio-economic inequalities in type 2 diabetes mellitus prevalence in Spain, 1987-2006. *Eur J Public Health*. 2012;22:765-771.

- (17) Muller G, Hartwig S, Greiser KH, et al. Gender differences in the association of individual social class and neighbourhood unemployment rate with prevalent type 2 diabetes mellitus: a cross-sectional study from the DIAB-CORE consortium. *BMJ Open.* 2013;3.
- (18) Tarlov AR. Public Policy Frameworks for Improving Population Health. *Ann N Y Acad Sci.* 2006;896:281-293.
- (19) Marmot MG, Shipley MJ. Do socioeconomic differences in mortality persist after retirement? 25 year follow up of civil servants from the first Whitehall study. *BMJ*. 1996;313:1177-1180.
- (20) Frieden TR. A framework for public health action: the health impact pyramid. *Am J Public Health*. 2010;100:590-595.
- (21) Fenton. Health Care's Blind Side: The Overlooked Connection between Social Needs and Good Health. Robert Wood Johnson Foundation; 2011.
- (22) Smedley, B. D., Stith, A. Y., and Nelson, A. R. Unequal treatment: confronting racial and ethnic disparities in health care. Smedley, B. D., Stith, A. Y., and Nelson, A. R. Institute of Medicine (US) Committee on Understanding and Eliminating Racial and Ethnic Disparities in Health Care . 2005. Washington, DC, National Academy Press.
- (23) Committee on the Recommended Social and Behavioral Domains and Measures for Electronic Health Records Board on Population Health and Public Health Practice. *Capturing Social and Behavioral Domains and Measures in Electronic Health Records PHASE 2*. Washington, DC: National Academies Press; 2014.
- (24) Centers for Disease Control and Prevention. CMS Timeline of Important MU Dates. http://www.cdc.gov/ehrmeaningfuluse/timeline.html . 2016. Accessed 9-9-2016.
- (25) Tagalicod, R. and Reider, J. Progress on Adoption of Electronic Health Records. https://www.cms.gov/eHealth/ListServ\_Stage3Implementation.html . 2016. Centers for Medicare & Medicaid Services. Accessed 9-12-2016.
- (26) HealthIT.gov. HITPC Meaningful Use Stage 3 Final Recommendations. https://www.healthit.gov/facas/sites/faca/files/HITPC\_MUWG\_Stage3\_Recs\_2014-04-01.pdf . 4-1-2014. Accessed 9-12-2016.
- (27) Centers for Medicare & Medicaid Services. MACRA: Delivery System Reform, Medicare Payment Reform. https://www.cms.gov/Medicare/Quality-Initiatives-Patient-Assessment-Instruments/Value-Based-Programs/MACRA-MIPS-and-APMs/MACRA-MIPS-and-APMs.html . 2016. Accessed 9-9-2016.
- (28) Centers for Medicare & Medicaid Services. CMS Quality Strategy 2016. https://www.cms.gov/medicare/quality-initiatives-patient-assessment-instruments/qualityinitiativesgeninfo/downloads/cms-quality-strategy.pdf . 2016. Accessed 9-9-2016.
- (29) The Office of the National Coordinator for Health Information Technology (ONC). Federal Health IT: Strategic Plan 2015-2020. https://www.healthit.gov/sites/default/files/9-5-federalhealthitstratplanfinal\_0.pdf. 2016. Office of the Secretary, United States Department of Health and Human Services. Accessed 10-17-2016.

- (30) The Menges Group. Positively Impacting Social Determinants of Health: How Safety Net Health Plans Lead the Way.

  <a href="http://www.communityplans.net/Portals/0/Fact%20Sheets/ACAP\_Plans\_and\_Social\_Determinants\_of\_Health.pdf">http://www.communityplans.net/Portals/0/Fact%20Sheets/ACAP\_Plans\_and\_Social\_Determinants\_of\_Health.pdf</a> . 2014. Accessed 9-12-2016.
- (31) Institute for Alternative Futures. Community Health Centers Leveraging the Social Determinants of Health. <a href="http://www.altfutures.org/pubs/leveragingSDH/IAF-CHCsLeveragingSDH.pdf">http://www.altfutures.org/pubs/leveragingSDH/IAF-CHCsLeveragingSDH.pdf</a> . 2012. Alexandria, VA. Accessed 9-12-2016.
- (32) Bachrach, D., Pfister, H., Wallis, K., and Lipson, M. Addressing Patients' Social Needs: An Emerging Business Case for Provider Investment, The Commonwealth Fund, The Skoll Foundation, and the Pershing Square Foundation. 5-29-2014.
- (33) Chung EK, Siegel BS, Garg A, et al. Screening for Social Determinants of Health Among Children and Families Living in Poverty: A Guide for Clinicians. *Curr Probl Pediatr Adolesc Health Care*. 2016;46:135-153.
- (34) Arvantes, James. Affordable Care Act Creates Greater Health Care Role for CHCs Number of Health Centers Expected to Double by 2015. <a href="http://www.aafp.org/news/government-medicine/20101117hcreformchcs.html">http://www.aafp.org/news/government-medicine/20101117hcreformchcs.html</a> . 2016. Accessed 10-17-2016.
- (35) National Association of Community Health Centers. The Safety Net on the Edge. NACHC. 2005. Bethesda, MD.
- (36) National Association of Community Health Centers. A Sketch Book of Community Health Centers: Chartbook 2014. http://www.nachc.com/client/Chartbook 2014.pdf . 2014. Accessed 9-28-2015.
- (37) Kaiser Family Foundation. Patients Served by Federally-Funded Federally Qualified Health Centers. <a href="http://kff.org/other/state-indicator/total-patients-served-by-fqhcs/">http://kff.org/other/state-indicator/total-patients-served-by-fqhcs/</a>. 2015. Accessed 10-6-2015.
- (38) Garg A, Jack B, Zuckerman B. Addressing the social determinants of health within the patient-centered medical home: lessons from pediatrics. *JAMA*. 2013;309:2001-2002.
- (39) Garg A, Toy S, Tripodis Y, Silverstein M, Freeman E. Addressing Social Determinants of Health at Well Child Care Visits: A Cluster RCT. *Pediatrics*. 2015;135:e296-e304.
- (40) Garg A, Sarkar S, Marino M, Onie R, Solomon BS. Linking urban families to community resources in the context of pediatric primary care. *Patient Educ Couns.* 2010;79:251-254.
- (41) Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. *Pediatrics*. 2007;120:547-558.
- (42) Page-Reeves J, Kaufman W, Bleecker M, et al. Addressing Social Determinants of Health in a Clinic Setting: The WellRx Pilot in Albuquerque, New Mexico. *J Am Board Fam Med.* 2016;29:414-418.
- (43) Matthews KA, Adler NE, Forrest CB, Stead WW. Collecting psychosocial "vital signs" in electronic health records: Why now? What are they? What's new for psychology? *Am Psychol.* 2016;71:497-504.
- (44) Giuse NB, Koonce TY, Kusnoor SV, et al. Institute of Medicine Measures of Social and Behavioral Determinants of Health: A Feasibility Study. *Am J Prev Med.* 2016.

- (45) Bodenheimer T, Ghorob A, Willard-Grace R, Grumbach K. The 10 building blocks of high-performing primary care. *Ann Fam Med.* 2014;12:166-171.
- (46) World Health Organization. What are social determinants of health? <a href="http://www.who.int/social\_determinants/sdh\_definition/en/">http://www.who.int/social\_determinants/sdh\_definition/en/</a>. 2-5-2016. Accessed 10-3-0016.
- (47) Williams DR, Costa MV, Odunlami AO, Mohammed SA. Moving upstream: how interventions that address the social determinants of health can improve health and reduce disparities. *J Public Health Manag Pract.* 2008;14 Suppl:S8-17.
- (48) Carter-Pokras O, Bereknyei S, Lie D, Braddock CH, III. Surmounting the unique challenges in health disparities education: a multi-institution qualitative study. *J Gen Intern Med.* 2010;25 Suppl 2:S108-S114.
- (49) National Research Council (US) and Institute of Medicine (US). U.S. Health in International Perspective: Shorter Lives, Poorer Health. 2013.
- (50) Levine DA, Allison JJ, Cherrington A, Richman J, Scarinci IC, Houston TK. Disparities in self-monitoring of blood glucose among low-income ethnic minority populations with diabetes, United States. *Ethn Dis.* 2009;19:97-103.
- (51) Robbins JM, Thatcher GE, Webb DA, Valdmanis VG. Nutritionist visits, diabetes classes, and hospitalization rates and charges: the Urban Diabetes Study. *Diabetes Care*. 2008;31:655-660.
- (52) Rhee MK, Cook CB, El-Kebbi I, et al. Barriers to diabetes education in urban patients: perceptions, patterns, and associated factors. *Diabetes Educ.* 2005;31:410-417.
- (53) Vest BM, Kahn LS, Danzo A, et al. Diabetes self-management in a low-income population: impacts of social support and relationships with the health care system. *Chronic Illn.* 2013;9:145-155.
- (54) Wallia A, Molitch ME. Insulin therapy for type 2 diabetes mellitus. JAMA. 2014;311:2315-2325.
- (55) Funnell MM, Anderson RM. MSJAMA: the problem with compliance in diabetes. JAMA. 2000;284:1709.
- (56) Russell LB, Suh DC, Safford MA. Time requirements for diabetes self-management: too much for many? *J Fam Pract*. 2005;54:52-56.
- (57) Jones-Smith JC, Karter AJ, Warton EM, et al. Obesity and the food environment: income and ethnicity differences among people with diabetes: the Diabetes Study of Northern California (DISTANCE). *Diabetes Care*. 2013;36:2697-2705.
- (58) Stoddard PJ, Laraia BA, Warton EM, et al. Neighborhood deprivation and change in BMI among adults with type 2 diabetes: the Diabetes Study of Northern California (DISTANCE). *Diabetes Care*. 2013;36:1200-1208.
- (59) Laraia BA, Karter AJ, Warton EM, Schillinger D, Moffet HH, Adler N. Place matters: neighborhood deprivation and cardiometabolic risk factors in the Diabetes Study of Northern California (DISTANCE). *Soc Sci Med.* 2012;74:1082-1090.
- (60) Zhang X, Geiss LS, Cheng YJ, Beckles GL, Gregg EW, Kahn HS. The missed patient with diabetes: how access to health care affects the detection of diabetes. *Diabetes Care*. 2008;31:1748-1753.

- (61) Lee HA, Lee KE, Jeong YW, et al. How do life-course trajectories of socioeconomic position affect quality of life in patients with diabetes mellitus? *Qual Life Res.* 2014;23:1337-1344.
- (62) Anekwe TD, Rahkovsky I. The association between food prices and the blood glucose level of US adults with type 2 diabetes. *Am J Public Health*. 2014;104:678-685.
- (63) Muennig P, Franks P, Jia H, Lubetkin E, Gold MR. The income-associated burden of disease in the United States. *Soc Sci Med.* 2005;61:2018-2026.
- (64) Keller D, Jones N, Savageau JA, Cashman SB. Development of a brief questionnaire to identify families in need of legal advocacy to improve child health. *Ambul Pediatr*. 2008;8:266-269.
- (65) Gottlieb L, Hessler D, Long D, Amaya A, Adler N. A randomized trial on screening for social determinants of health: the iScreen study. *Pediatrics*. 2014;134:e1611-e1618.
- (66) Gottlieb, L. Social Needs Screening and Interventions at CHO and SFGH: Results from the iScreen and Pediatrics Help Desks Studies. Presentation at Bay Area Research Consortium on Toxic Stress and Health. 2015. 9-29-2014.
- (67) Silverstein M, Conroy K, Sandel M. Screening for social determinants of health in pediatric primary care. *Pediatr Ann.* 2008;37:740-746.
- (68) Walker RJ, Smalls BL, Campbell JA, Strom Williams JL, Egede LE. Impact of social determinants of health on outcomes for type 2 diabetes: a systematic review. *Endocrine*. 2014;47:29-48.
- (69) Whiting D, Unwin N, Roglic G. Diabetes: equity and social determinants. *Equity, social determinants and public health programmes*. Geneva: World Health Organization; 2010:77-94.
- (70) Maddigan SL, Feeny DH, Majumdar SR, Farris KB, Johnson JA. Understanding the determinants of health for people with type 2 diabetes. *Am J Public Health*. 2006;96:1649-1655.
- (71) Liburd LC, Jack L, Jr., Williams S, Tucker P. Intervening on the social determinants of cardiovascular disease and diabetes. *Am J Prev Med.* 2005;29:18-24.
- (72) Dubowitz T, Heron M, Bird CE, et al. Neighborhood socioeconomic status and fruit and vegetable intake among whites, blacks, and Mexican Americans in the United States. *Am J Clin Nutr.* 2008;87:1883-1891.
- (73) James WP, Nelson M, Ralph A, Leather S. Socioeconomic determinants of health. The contribution of nutrition to inequalities in health. *BMJ*. 1997;314:1545-1549.
- (74) Roos G, Johansson L, Kasmel A, Klumbiene J, Prattala R. Disparities in vegetable and fruit consumption: European cases from the north to the south. *Public Health Nutr.* 2001;4:35-43.
- (75) Capon AG. Health impacts of urban development: key considerations. *N S W Public Health Bull.* 2007;18:155-156.
- (76) Knowler WC, Barrett-Connor E, Fowler SE, et al. Reduction in the incidence of type 2 diabetes with life-style intervention or metformin. *N Engl J Med.* 2002;346:393-403.
- (77) Tuomilehto J, Eriksson JG, Valle TT, et al. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. *N Engl J Med.* 2001;344:1343-1350.

- (78) Brown AF, Ettner SL, Piette J, et al. Socioeconomic position and health among persons with diabetes mellitus: a conceptual framework and review of the literature. *Epidemiol Rev.* 2004;26:63-77.
- (79) Office of Disease Prevention and Health Promotion. Healthy People 2020.
  <a href="http://www.healthypeople.gov/">http://www.healthypeople.gov/</a>. 2015. U.S. Department of Health and Human Services. Accessed 9-28-2015.
- (80) Gottlieb LM, Tirozzi KJ, Manchanda R, Burns AR, Sandel MT. Moving electronic medical records upstream: Incorporating social determinants of health. *Am J Prev Med.* 2015;48.
- (81) Pinto AD, Glattstein-Young G, Mohamed A, Bloch G, Leung FH, Glazier RH. Building a Foundation to Reduce Health Inequities: Routine Collection of Sociodemographic Data in Primary Care. *J Am Board Fam Med.* 2016;29:348-355.
- (82) Alley DE, Asomugha CN, Conway PH, Sanghavi DM. Accountable Health Communities--Addressing Social Needs through Medicare and Medicaid. *N Engl J Med.* 2016;374:8-11.
- (83) Health and Human Services Department. 2015 Edition Health Information Technology (Health IT) Certification Criteria, 2015 Edition Base Electronic Health Record (EHR) Definition, and ONC Health IT Certification Program Modifications. https://www.federalregister.gov/articles/2015/03/30/2015-06612/2015-edition-health-information-technology-health-it-certification-criteria-2015-edition-base#p-1748 . 2016. Accessed 9-28-2016.
- (84) Stringhini S, Batty GD, Bovet P, et al. Association of lifecourse socioeconomic status with chronic inflammation and type 2 diabetes risk: the Whitehall II prospective cohort study. *PLoS Med.* 2013;10:e1001479.
- (85) Gottlieb LM, Hessler D, Long D, et al. Effects of Social Needs Screening and In-Person Service Navigation on Child Health: A Randomized Clinical Trial. *JAMA Pediatr.* 2016;e162521.
- (86) De Vito Dabbs A, Myers BA, Mc Curry KR, et al. User-centered design and interactive health technologies for patients. *Comput Inform Nurs.* 2009;27:175-183.
- (87) Henderson VA, Barr KL, An LC, et al. Community-based participatory research and user-centered design in a diabetes medication information and decision tool. *Prog Community Health Partnersh.* 2013;7:171-184.
- (88) LeRouge C, Wickramasinghe N. A review of user-centered design for diabetes-related consumer health informatics technologies. *J Diabetes Sci Technol.* 2013;7:1039-1056.
- (89) Steele GC, Khan AI, Kuluski K, et al. Improving Patient Experience and Primary Care Quality for Patients With Complex Chronic Disease Using the Electronic Patient-Reported Outcomes Tool: Adopting Qualitative Methods Into a User-Centered Design Approach. *JMIR Res Protoc.* 2016;5:e28.
- (90) Witteman HO, Dansokho SC, Colquhoun H, et al. User-centered design and the development of patient decision aids: protocol for a systematic review. *Syst Rev.* 2015;4:11.
- (91) Cooper RG. Overhauling the New Product Process. Journal of Consumer Research. 1996;25:482.

- (92) Rauterberg M, Strohm O. Benefits of user-oriented software development based on an iterative cyclic process model for simultaneous engineering. *International Journal of Industrial Ergonomics*. 1995;16:391-410.
- (93) Schleyer TK, Thyvalikakath TP, Hong J. What is user-centered design? *J Am Dent Assoc.* 2007;138:1081-1082.
- (94) DeVoe JE, Bazemore AW, Cottrell EK, et al. Perspectives in Primary Care: A Conceptual Framework and Path for Integrating Social Determinants of Health Into Primary Care Practice. *Ann Fam Med*. 2016;14:104-108.
- (95) Powell BJ, McMillen JC, Proctor EK, et al. A compilation of strategies for implementing clinical innovations in health and mental health. *Med Care Res Rev.* 2012;69:123-157.
- (96) Powell BJ, Waltz TJ, Chinman MJ, et al. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. *Implement Sci.* 2015;10:21.
- (97) Powell BJ, Beidas RS, Lewis CC, et al. Methods to Improve the Selection and Tailoring of Implementation Strategies. *J Behav Health Serv Res.* 2015.
- (98) Proctor EK, Powell BJ, McMillen JC. Implementation strategies: recommendations for specifying and reporting. *Implement Sci.* 2013;8:139.
- (99) Godley SH, Garner BR, Smith JE, Meyers RJ, Godley MD. A large-scale dissemination and implementation model for evidence-based treatment and continuing care. *Clin Psychol (New York)*. 2011;18:67-83.
- (100) Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. *Milbank Q.* 2004;82:581-629.
- (101) Massoud, M. R., Nielson, G. A., Nolan, K., Schall, M. W., and Sevin, C. A Framework for Spread: From Local Improvements to System-Wide Change. IHI Innovation Series white paper. Cambridge, MA: Institute for Healthcare Improvement. <a href="https://www.IHI.org">www.IHI.org</a>. 2006. 1-8-2013.
- (102) Paina L, Peters DH. Understanding pathways for scaling up health services through the lens of complex adaptive systems. *Health Policy Plan.* 2012;27:365-373.
- (103) Lukas CV, Meterko MM, Mohr D, et al. Implementation of a clinical innovation: the case of advanced clinic access in the Department of Veterans Affairs. *J Ambul Care Manage*. 2008;31:94-108.
- (104) Solberg LI. Improving medical practice: a conceptual framework. Ann Fam Med. 2007;5:251-256.
- (105) Janovsky, K., Peters, D. H., Arur, A., and Sundaram, S. Improving health services and strengthening health systems: adopting and implementing innovative strategies. Making Health Systems Work, Working Paper No. 5. Geneva: World Health Organization, Evidence and Information for Policy. 2006.
- (106) Taylor EF, Machta RM, Meyers DS, Genevro J, Peikes DN. Enhancing the primary care team to provide redesigned care: the roles of practice facilitators and care managers. *Ann Fam Med.* 2013;11:80-83.
- (107) Munoz M, Pronovost P, Dintzis J, et al. Implementing and evaluating a multicomponent inpatient diabetes management program: putting research into practice. *Jt Comm J Qual Patient Saf.* 2012;38:195-206.

- (108) Weir C, McLeskey N, Brunker C, Brooks D, Supiano MA. The role of information technology in translating educational interventions into practice: an analysis using the PRECEDE/PROCEED model. *J Am Med Inform Assoc.* 2011;18:827-834.
- (109) Office of the National Coordinator for Health Information Technology. 2015 Edition §170.315(a)(15) Social, Psychological, and Behavioral Data. https://www.healthit.gov/sites/default/files/170\_315a15\_social\_behavioral\_data\_v10.pdf . 2016. Accessed 9-28-2016.
- (110) DeVoe JE, Gold R, McIntire P, Puro J, Chauvie S, Gallia CA. Electronic health records vs Medicaid claims: completeness of diabetes preventive care data in community health centers. *Ann Fam Med.* 2011;9:351-358.
- (111) DeVoe JE, Gold R, Cottrell E, et al. The ADVANCE network: accelerating data value across a national community health center network. *J Am Med Inform Assoc.* 2014;21:271-278.
- (112) OCHIN. Collaboration and Innovation through Research. https://ochin.org/ochin-research/ . 2016. Accessed 10-17-2016.
- (113) Gold R, Bunce A, Cohen DJ, DeVoe JE, Hollombe C, Nelson C. Reporting on implementation strategies: An example from an intervention adapted across care settings. *Ann Fam Med*. In press.
- (114) Gold R, Nelson C, Cowburn S, et al. Feasibility and Impact of Implementing a Private Care System's Diabetes Quality Improvement Intervention in the Safety Net: A Cluster-Randomized Trial. *Implementation Science*. 2015;10.
- (115) Gold R, Hollombe C, Bunce A, et al. Practices Enabling Implementation and Adaptation in the Safety Net (SPREAD-NET)': A pragmatic trial comparing implementation strategies. *Implementation Science*. 2015;10:144.
- (116) Lessard S, Bareil C, Lalonde L, et al. External facilitators and interprofessional facilitation teams: a qualitative study of their roles in supporting practice change. *Implement Sci.* 2016;11:97.
- (117) Chambers DA, Norton WE. The Adaptome: Advancing the Science of Intervention Adaptation. *Am J Prev Med.* 2016.
- (118) Maclean CD, Gagnon M, Callas P, Littenberg B. The Vermont diabetes information system: a cluster randomized trial of a population based decision support system. *J Gen Intern Med.* 2009;24:1303-1310.
- (119) Zai AH, Grant RW, Estey G, et al. Lessons from implementing a combined workflow-informatics system for diabetes management. *J Am Med Inform Assoc.* 2008;15:524-533.
- (120) Montori VM, Dinneen SF, Gorman CA, et al. The impact of planned care and a diabetes electronic management system on community-based diabetes care: the Mayo Health System Diabetes Translation Project. *Diabetes Care*. 2002;25:1952-1957.
- (121) Gottlieb L, Sandel M, Adler NE. Collecting and applying data on social determinants of health in health care settings. *JAMA Intern Med.* 2013;173:1017-1020.

- (122) Institute of Medicine. Recommended social and behavioral domains and measures for electronic health records. <a href="http://www.iom.edu/Activities/PublicHealth/SocialDeterminantsEHR.aspx">http://www.iom.edu/Activities/PublicHealth/SocialDeterminantsEHR.aspx</a> . 2014. National Academies of Science. 2-5-0216. Accessed 9-28-2016.
- (123) Garg AX, Adhikari NK, McDonald H, et al. Effects of computerized clinical decision support systems on practitioner performance and patient outcomes: a systematic review. *JAMA*. 2005;293:1223-1238.
- (124) Onie, R., Farmer, P., and Behforouz, H. Realigning Health with Care. http://www.ssireview.org/articles/entry/realigning health with care . 2012. 5-31-2014.
- (125) Health Resources & Services Administration, Bureau of Primary Health Care. Health Center Fact Sheet. http://bphc.hrsa.gov/about/healthcenterfactsheet.pdf . 2016. Accessed 9-28-2016.
- (126) Nichols GA, McBurnie M, Paul L, et al. The High Prevalence of Diabetes in a Large Cohort of Patients Drawn From Safety Net Clinics. *Prev Chronic Dis.* 2016;13:E78.
- (127) Blackwell DL, Lucas JW, Clarke TC. Summary health statistics for U.S. adults: National Health Interview Survey, 2012. National Center for Health Statistics. *Vital Health Stat.* 2014;10.
- (128) National Institute of Diabetes and Digestive and Kidney Diseases. Delaying or Preventing Type 2
  Diabetes. https://www.niddk.nih.gov/health-information/diabetes/delaying-preventing-type-2-diabetes
  . 2016. U.S. Department of Health and Human Services. Accessed 9-28-2016.
- (129) Division for Heart Disease and Stroke Prevention. Cholesterol Fact Sheet. http://www.cdc.gov/dhdsp/data\_statistics/fact\_sheets/docs/fs\_cholesterol.pdf . 2015. 9-17-2015.
- (130) Ali MK, Bullard KM, Saaddine JB, Cowie CC, Imperatore G, Gregg EW. Achievement of goals in U.S. diabetes care, 1999-2010. *N Engl J Med.* 2013;368:1613-1624.
- (131) Gold R, Nelson C, Cowburn S, et al. Feasibility and impact of implementing a private care system's diabetes quality improvement intervention in the safety net: a cluster-randomized trial. *Implement Sci.* 2015;10:83.
- (132) Casciato A, Angier H, Milano C, Gideonse N, Gold R, DeVoe JE. A practice-based approach to demonstrate the use of pediatric quality measures in outpatient electronic health record data. *Journal of the American Board of Family Medicine*. 2012;25:686-693.
- (133) Casciato A, Angier H, Milano C, Gideonse N, Gold R, DeVoe J. Are pediatric quality care measures too stringent? *J Am Board Fam Med.* 2012;25:686-693.
- (134) DeVoe JE, Tillotson CJ, Wallace LS, Angier H, Carlson MJ, Gold R. Parent and child usual source of care and children's receipt of health care services. *Ann Fam Med.* 2011;9:504-513.
- (135) DeVoe JE, Gold R, Spofford M, et al. Developing a network of community health centers with a common electronic health record: description of the Safety Net West Practice-based Research Network (SNW-PBRN). *J Am Board Fam Med.* 2011;24:597-604.
- (136) Angier, H., Wiggins, N., Gregg, J., Gold, R., and DeVoe, J. E. Engagement of Community Health Workers In a Health Policy Research Project Through a Novel Technique: The Community Retreat Paper presented at: North American Primary Care Research Group 2011; Banff, Alberta. 2011.

- (137) Gold R, Whitlock EP, Patnode CD, McGinnis PS, Buckley DI, Morris C. Prioritizing research needs based on a systematic evidence review: a pilot process for engaging stakeholders. *Health Expect.* 2011;doi: 10.1111/j.1369-7625.2011.00716.x. [Epub ahead of print].
- (138) Gold R, Angier H, Mangione-Smith R, et al. Feasibility of evaluating the CHIPRA care quality measures in electronic health record data. *Pediatrics*. 2012;130:139-149.
- (139) Gold, R., Meunch, J., Hill.C., Milano, C., Turner, A., Nelson, C., Mital, M., DeVoe, J., and Puro, J. Can a Privately Developed Quality Improvement Initiative be Adapted for Implementation in Primary Care Safety Net Clinics? Oral presentation: December 2012 at the 40th Annual North American Primary Care Research Group conference. New Orleans, LA. 12-5-2012. 12-5-2012.
- (140) Gold R, Connell FA, Heagerty P, Bezruchka S, Davis R, Cawthon ML. Income inequality and pregnancy spacing. *Soc Sci Med.* 2004;59:1117-1126.
- (141) Gold R, Kawachi I, Kennedy BP, Lynch JW, Connell FA. Ecological analysis of teen birth rates: association with community income and income inequality. *Matern Child Health J.* 2001;5:161-167.
- (142) Gold R, Kennedy B, Connell F, Kawachi I. Teen births, income inequality, and social capital: developing an understanding of the causal pathway. *Health Place*. 2002;8:77-83.
- (143) Gold R, Connell FA, Heagerty P, et al. Predicting time to subsequent pregnancy. *Matern Child Health J.* 2005;9:219-228.
- (144) National Institutes of Health. Training Institute for Dissemination and Implementation Research in Health 2012. 6-5-2012.
- (145) Gold R, Muench J, Hill C, et al. Collaborative development of a randomized study to adapt a diabetes quality improvement initiative for federally qualified health centers. *J Health Care Poor Underserved*. 2012;23:236-246.
- (146) Gold, R., Nichols, G, Muench, J, Hill, C, Mital, M, Dudl, J, DeVoe, J, Puro, J, and Nelson, C. Implementing an Integrated Care Setting's Diabetes QI Initiative in Safety Net Clinics: A Practice-Based Randomized Trial. Oral presentation: March 2012 at the 5<sup>th</sup> Annual NIH conference on the Science of Dissemination and implementation: Science at the Crossroads. Bethesda, MD. 3-20-2012.
- (147) DeVoe J, Angier H, Likumahuwa S, et al. Use of qualitative methods and user-centered design to develop customized health information technology tools within federally qualified health centers to keep children insured. *J Ambul Care Manage*. 2014;37:148-154.
- (148) DeVoe JE, Angier H, Burdick T, Gold R. Health information technology: an untapped resource to help keep patients insured. *Ann Fam Med.* 2014;12:568-572.
- (149) Gold R, Nelson C, Cowburn S, et al. Feasibility and Impact of Implementing a Private Care System's Diabetes Quality Improvement Intervention in the Safety Net: A Cluster-Randomized Trial. *Implementation Science*. 2015;10.
- (150) Angier H, Marino M, Sumic A, et al. Innovative Methods for Parents And Clinics to Create Tools for Kids' Care (IMPACCT Kids' Care) Study Protocol. *Contemp Clin Trials*. 2015.

- (151) DeVoe JE, Hoopes M, Nelson CA, et al. Impact of Electronic Health Record Tools on Children's Insurance Coverage: A Mixed Methods Study (Submitted May 2016). *Pediatrics*. 2016.
- (152) Lau R, Stevenson F, Ong BN, et al. Achieving change in primary care--effectiveness of strategies for improving implementation of complex interventions: systematic review of reviews. BMJ Open. 2015;5:e009993.
- (153) Thorpe KE, Zwarenstein M, Oxman AD, et al. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. *J Clin Epidemiol*. 2009;62:464-475.
- (154) Patsopoulos NA. A pragmatic view on pragmatic trials. Dialogues Clin Neurosci. 2011;13:217-224.
- (155) Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. *JAMA*. 2003;290:1624-1632.
- (156) NCQA. PCMH Eligility. http://www.ncqa.org/about-ncqa/contact-us. 2016. Accessed 9-28-2016.
- (157) Pawson R, Tilley N. Realistic Evaluation. London: SAGE Publications; 1997.
- (158) Dalkin SM, Greenhalgh J, Jones D, Cunningham B, Lhussier M. What's in a mechanism? Development of a key concept in realist evaluation. *Implement Sci.* 2015;10:49.
- (159) Lacouture A, Breton E, Guichard A, Ridde V. The concept of mechanism from a realist approach: a scoping review to facilitate its operationalization in public health program evaluation. *Implement Sci.* 2015;10:153.
- (160) Moore GF, Audrey S, Barker M, et al. Process evaluation of complex interventions: Medical Research Council guidance. *BMJ*. 2015;350:h1258.
- (161) Van Belle S, Wong G, Westhorp G, et al. Can "realist" randomised controlled trials be genuinely realist? *Trials*. 2016;17:313.
- (162) Marchal B, Westhorp G, Wong G, et al. Realist RCTs of complex interventions an oxymoron. *Soc Sci Med.* 2013;94:124-128.
- (163) McHugh S, Tracey ML, Riordan F, O'Neill K, Mays N, Kearney PM. Evaluating the implementation of a national clinical programme for diabetes to standardise and improve services: a realist evaluation protocol. *Implement Sci.* 2016;11:107.
- (164) Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. *Contemp Clin Trials*. 2007;28:182-191.
- (165) Coronado GD, Vollmer WM, Petrik A, et al. Strategies and opportunities to STOP colon cancer in priority populations: pragmatic pilot study design and outcomes. *BMC Cancer*. 2014;14:55.
- (166) Coronado GD, Burdick T, Petrik A, Kapka T, Retecki S, Green B. Using an Automated Data-driven, EHR-Embedded Program for Mailing FIT kits: Lessons from the STOP CRC Pilot Study. *J Gen Pract.* 2014;2:doi: 10.4172/2329-9126.1000141.
- (167) Coronado GD, Sanchez J, Petrik A, Kapka T, DeVoe J, Green B. Advantages of wordless instructions on how to complete a fecal immunochemical test: lessons from patient advisory council members of a federally qualified health center. *J Cancer Educ.* 2014;29:86-90.

- (168) Coronado GD, Petrik A, Spofford M, et al. Perceptions of under and overutilization of cervical cancer screening services at Latino-serving community health centers. *J Community Health*. 2013;38:915-918.
- (169) Bailey SR, O'Malley JP, Gold R, Heintzman J, Likumahuwa S, DeVoe JE. Diabetes care quality is highly correlated with patient panel characteristics. *J Am Board Fam Med*. 2013;26:669-679.
- (170) Dean CB, Nielsen JD. Generalized linear mixed models: a review and some extensions. *Lifetime Data Anal.* 2007;13:497-512.
- (171) UCSF Center for Excellence in Primary Care. Building Blocks of Primary Care Assessment (BBPCA). https://cepc.ucsf.edu/sites/cepc.ucsf.edu/files/Building%20Blocks%20Assessment.pdf . 2016. Accessed 9-28-2016.
- (172) Chinman M, Acosta J, Ebener P, Malone PS, Slaughter ME. Can implementation support help community-based settings better deliver evidence-based sexual health promotion programs? A randomized trial of Getting To Outcomes(R). *Implement Sci.* 2016;11:78.
- (173) Frieden TR. Forward: CDC Health Disparities and Inequalities Report United States, 2011. *MMWR Surveill Summ.* 2011;60 Suppl:1-2.
- (174) Barnett E, Casper M. A definition of "social environment". Am J Public Health. 2001;91:465.
- (175) Palloni A, Palloni G. Education, earnings, and diabetes. Health Aff (Millwood). 2012;31:1126.
- (176) van Lenthe FJ, Borrell LN, Costa G, et al. Neighbourhood unemployment and all cause mortality: a comparison of six countries. *J Epidemiol Community Health*. 2005;59:231-237.
- (177) Puig-Barrachina V, Malmusi D, Martenez JM, Benach J. Monitoring social determinants of health inequalities: the impact of unemployment among vulnerable groups. *Int J Health Serv.* 2011;41:459-482.
- (178) Mete C. Predictors of elderly mortality: health status, socioeconomic characteristics and social determinants of health. *Health Econ.* 2005;14:135-148.
- (179) McCarthy M. Social determinants and inequalities in urban health. Rev Environ Health. 2000;15:97-108.
- (180) Marmot M. Social determinants of health inequalities. Lancet. 2005;365:1099-1104.
- (181) Kreatsoulas C, Anand SS. The impact of social determinants on cardiovascular disease. *Can J Cardiol.* 2010;26 Suppl C:8C-13C.
- (182) Gold R, Bunce AE, Cohen DJ, et al. Reporting on the strategies needed to implement proven interventions: An example from a "real-world" cross-setting implementation study. *Mayo Clin Proc.* 2016.
- (183) Olson R, Thompson SV, Elliot DL, et al. Safety and Health Support for Home Care Workers: The COMPASS Randomized Controlled Trial. *Am J Public Health*. 2016;106:1823-1832.
- (184) Marino M, Killerby M, Lee S, et al. The effects of a cluster randomized controlled workplace intervention on sleep and work-family conflict outcomes in an extended care setting. Sleep Health: Journal of the National Sleep Foundation.

- (185) Melnick AL, Rdesinski RE, Marino M, et al. Randomized Controlled Trial of Home-Based Hormonal Contraceptive Dispensing for Women At Risk of Unintended Pregnancy. *Perspect Sex Reprod Health*. 2016;48:93-99.
- (186) Rothman KJ. No adjustments are needed for multiple comparisons. Epidemiology. 1990;1:43-46.
- (187) Perneger TV. What's wrong with Bonferroni adjustments. BMJ. 1998;316:1236-1238.
- (188) Xu Z, Kalbfleisch JD. Propensity score matching in randomized clinical trials. *Biometrics*. 2010;66:813-823.
- (189) Little RJ, Rubin DB. Causal effects in clinical and epidemiological studies via potential outcomes: concepts and analytical approaches. *Annu Rev Public Health*. 2000;21:121-145.
- (190) Hayes RJ, Alexander ND, Bennett S, Cousens SN. Design and analysis issues in cluster-randomized trials of interventions against infectious diseases. *Stat Methods Med Res.* 2000;9:95-116.
- (191) Schierhout G, Hains J, Si D, et al. Evaluating the effectiveness of a multifaceted, multilevel continuous quality improvement program in primary health care: developing a realist theory of change. *Implement Sci.* 2013;8:119.
- (192) Lewis JH, Whelihan K, Navarro I, Boyle KR. Community health center provider ability to identify, treat and account for the social determinants of health: a card study. *BMC Fam Pract.* 2016;17:121.
- (193) Westfall JM, Zittleman L, Ringel M, et al. How do rural patients benefit from the patient-centred medical home? A card study in the High Plains Research Network. *London J Prim Care (Abingdon ).* 2014;6:136-148.
- (194) Fetters MD, Curry LA, Creswell JW. Achieving integration in mixed methods designs-principles and practices. *Health Serv Res.* 2013;48:2134-2156.
- (195) Powell BJ, Proctor EK, Glisson CA, et al. A mixed methods multiple case study of implementation as usual in children's social service organizations: study protocol. *Implement Sci.* 2013;8:92.
- (196) Glaser BG, Strauss AL. *The discovery of grounded theory: Strategies for qualitative research*. New York: Aldine de Gruyter; 1999.
- (197) Strauss A, Corbin J. *Basics of qualitative research: Techniques and procedures for developing grounded theory (2<sup>nd</sup> ed.)*. Thousand Oaks, CA: Sage; 1998.
- (198) Charmaz K. Grounded Theory Methods in Social Justice Research. In: Denzin NK, Lincoln YS, eds. *The SAGE Handbook of Qualitative Research*, 4<sup>th</sup> ed. Thousand Oaks, CA: Sage Publications, Inc.; 2011:359-80.
- (199) Borkan J. Immersion/crystallization. In: Crabtree BF, Miller WL, eds. *Doing qualitative research*. 2nd ed ed. Thousand Oaks, CA: Sage Publications, Inc.; 1999:179-94.
- (200) Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. *Health Serv Res.* 2007;42:1758-1772.
- (201) Byng R, Norman I, Redfern S, Jones R. Exposing the key functions of a complex intervention for shared care in mental health: case study of a process evaluation. *BMC Health Serv Res.* 2008;8:274.

- (202) Little, T. D., Schnabel, K. U., and Baumert, J. Modeling longitudinal and multilevel data: Practical issues, applied approaches, and specifc examples. 2000. Mahwah, NJ, Erlbaum.
- (203) Little RJA, Rubin DB. *Introduction, in Statistical Analysis with Missing Data, Second Edition*. Hoboken, NJ, USA: John Wiley & Sons, Inc.; 2002.
- (204) Schafer JL. Analysis of Incomplete Multivariate Data. London, UK: Chapman & Hall/CRC Press; 1997.